CLINICAL TRIAL: NCT05294796
Title: Efficacy and Safety of Different Antimicrobial Durations for the Treatment of Infections Associated With Osteosynthesis Material Implanted After Long Bone Fractures (DURATIOM). Phase 3 Pragmatic Multicenter Open Labelled Randomized Trial.
Brief Title: Efficacy and Safety of Antimicrobial Durations Treatment of Infections Associated With Osteosynthesis Material
Acronym: DURATIOM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DURATIOM
Record Dates: First submitted 2022-01-26; First posted 2022-03-24 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-03

CONDITIONS: Infections
Keywords: Infections associated with osteosynthesis material; Fracture-related infection; Long bone fractures; Antibiotics duration; Antimicrobial therapy; Multidrug-resistant bacteria; Biofilm fracture healing; Antibiotic toxicity; Investigator-driven clinical trial
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Pragmatic, multicenter, non-inferiority, open labelled, randomized trial comparing different durations of antibiotherapy in osteosynthesis material infections after long bone fractures treated with debridement and material retention (see design algorithm and inclusion criteria). The CONSORT extension for pragmatic designs will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short course of antibiotherapy (Active Comparator): Patients enrolled in this arm, will receive 8 weeks of antibiotherapy in case of early infection (< 2 week), and 12 weeks of antibiotherapy in case of delayed infection (2-10 weeks)
  Interventions: Combination Product: Short course of antibiotherapy
- Long course of antibiotherapy (Active Comparator): Patients enrolled in this arm, will receive 12 weeks of antibiotherapy in case of early infection (< 2 week), and until fracture healing of antibiotherapy in case of delayed infection
  Interventions: Combination Product: Long course of antibiotherapy

INTERVENTIONS:
Combination Product: Short course of antibiotherapy — Short duration of authorized antibiotic therapy according to its data sheet in infections associated with osteosynthesis material
  Arms: Short course of antibiotherapy
Combination Product: Long course of antibiotherapy — Long duration of authorized antibiotic therapy according to its data sheet in infections associated with osteosynthesis material
  Arms: Long course of antibiotherapy

SUMMARY:
Infections associated with osteosynthesis material are among the most feared and challenging complications of trauma surgery and can lead to total function loss or limb amputation when complete recovery is to be expected without infection.

This is a clinical trial with the purpose of evaluate the optimal duration of antibiotic therapy in Infections Associated With Osteosynthesis Material Implanted when implant is retained.

DETAILED DESCRIPTION:
Orthopedic implants for fracture fixation or osteosynthesis material are used for internal fixation of fractures, allowing their stability and consolidation.

Infection associated with osteosynthesis material is one of the most feared and challenging complications of trauma surgery and can lead to total loss of function or amputation of the limb, when complete recovery is to be expected without infection. Furthermore, they involve excessive consumption of antimicrobials, with inadequate prescriptions and prolonged durations that favour superinfections by multidrug-resistant microorganisms, in addition to the drug-related toxicities, especially diarrhea due to Clostridium difficile. Most studies and recommendations on the management of orthopedic implant-associated infections have focused on prosthetic joint infections, and while they share similarities with Infections Associated With Osteosynthesis Material Implanted, there are major differences in terms of risk factors, diagnosis, treatment, and prevention. While the extrapolation of knowledge from prosthetic joint infections to the field of Infections Associated With Osteosynthesis Material Implanted has helped orthopedic surgeons and internists/infectologists in their management, there are large gaps and unanswered questions that represent a new challenge for research in this field. One of these challenges, and focusing on the field of infection treatment, is the search for the best surgical procedure according to the age of the implant and fracture healing, to determine the duration of antibiotic treatment and whether it should be maintained until fracture healing, and which is the most appropriate treatment in each of the scenarios.

The identification of conditions in which the duration of the antimicrobial treatment can be shortened, and in case of prolonged treatments, which antimicrobial has the best safety profile and less impact on the induction of bacterial resistances is of special interest, due to the frequent appearance of toxicities and the increase of bacterial resistances and superinfections by multidrug-resistant bacteria.

If the hypothesis of non-inferiority of short vs. long antibiotic treatments is demonstrated, and the efficacy of antibiotics with less ecological impact in long treatments, the impact on reduction of bacterial resistance, toxicity and health costs will be observed. The project also aims to promote quality and multidisciplinary care, homogenising clinical practice in the management of Infections Associated With Osteosynthesis Material Implanted based on scientific knowledge. Early and personalised patient care with Infections Associated With Osteosynthesis Material Implanted allows for faster recovery, both clinically and functionally, enabling earlier mobility recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 14 years.
* Stable fracture, even if unconsolidated.
* Controlled infection (absence of signs or symptoms of sepsis).
* Early or delayed infection.
* Availability of antibiotics active against the isolated microorganism.
* Absence of bone exposure. Patients who initially had bone exposure but during the debridement surgery bone coverage was performed by any method (skin approximation, grafting, vacuum therapy) can be included in the criteria.
* Signed written informed consent.
* If there is a possibility of pregnancy (in women of childbearing potential) or paternity, agree to use a highly effective method of birth control recommended by the Clinical Trial Facilitation Group (CTFG) during the treatment phase of the trial

Exclusion Criteria:

* Late infections
* Infections of osteosynthesis material in non-long bones.
* Infections of revision osteosynthesis material or occurring after previous surgeries.
* Patients who are not expected to be followed up for at least 1 year after completion of antibiotic treatment.
* Pregnant or lactating women.
* Patients in whom there may be drug interactions or contraindications described in the technical data sheets of the investigational drugs used in this trial.
* Infections due to mycobacteria, fungi and parasites (since they are infections that are treated with drugs and for different durations).
* Patients in whom all the material is replaced during the debridement at the same surgical time (since these patients require antibiotic treatment for less than 8 weeks in all cases).
* Infections of external fixators.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinical cure in the test of cure | 12 months after completion of antimicrobial treatment
  A success at the test of cure is the resolution of infection symptoms, the absence of clinical signs and symptoms of infection (persistence of symptoms of infection, relapse of infection after a period without symptoms, or superinfection by a different microorganism) without antibiotic therapy and with C-reactive protein <10 mg/L (unless another cause justifies a higher C-reactive protein value); If the patient dies, when the death was not related to the infection; and no need for chronic suppressive antibiotic therapy to "control" of the infection.
Radiological healing in the test of cure | 12 months after completion of antimicrobial treatment
  Radiological healing is defined as the presence of radiological signs of fracture consolidation (plain radiographic or CT) of the infected bone. Non-union or absence of consolidation of a fractured bone is defined when it has not completely healed within 9 months after osteosynthesis surgery or when it has not shown progression towards fracture callus formation in 3 consecutive months on serial radiographs.
  The REBORNE fracture healing scale will be used for a more accurate assessment of fracture healing on radiographs, or CT if necessary.
Definitive soft tissue coverage at test of cure | 12 months after completion of antimicrobial treatment
  Number of patients who present definitive soft tissue coverage at test of cure

SECONDARY OUTCOMES:
Efficacy of each group of antibiotics | 12 months from the start of antibiotic treatment
  Number of days of antibiotic administration
Performance of an antibiogram to assess the development of antimicrobial resistance | 8 months and 12 months
  Standard microbiological techniques will be used to identify microorganisms recovered and to determine antimicrobial susceptibility according to EUCAST recommendation (EUCAST guidelines for detection of resistance mechanisms and specific resistances of clinical and/or epidemiological importance, Version 2.0, 2017) https://www.eucast.org/fileadmin/src/media/PDFs/EUCAST_files/Resistance_mechanisms/EUCAST_detection_of_resistance_mechanisms_170711.pdf
Surgical wound culture to assess the development of secondary infections | 8 months and 12 months
  To evaluate the appearance of secondary infections during antibiotic treatment that standard microbiological techniques will be used to identify microorganisms recovered and to determine antimicrobial susceptibility according to EUCAST recommendation (EUCAST guidelines for detection of resistance mechanisms and specific resistances of clinical and/or epidemiological importance, Version 2.0, 2017) https://www.eucast.org/fileadmin/src/media/PDFs/EUCAST_files/Resistance_mechanisms/EUCAST_detection_of_resistance_mechanisms_170711.pdf
Recurrence rate | 8 months and 12 months
  To evaluate the recurrence rate during antibiotic treatment.
Evaluate the need for new surgeries, such as debridement, removal of material, coverage or amputation, through radiological evaluation of fracture union. | Day 28, week 8, week 12, month 6 and month 12.
  To evaluate the need for new surgeries through radiological evaluation
Evaluation of the functional status, defined as the recovery of the functionality of the limb prior to the fracture, by completing the Quick Disabilities of Arm, Shoulder and Hand questionnaire. | 6 months and 12 months (visit 6 and 7)
  The functional state, normal or reduced, will be evaluated with respect to the situation prior to the fracture. Lower extremity mobility is classified as: walks unassisted; with 1 cane; with 2 canes; with walker; "wander home alone"; not wandering..
Evaluation the consumption of health resources | Month 12
  Total number and posology of all the antibiotics that have been administered to the patient will be taken into account, in addition to the new surgeries, new microbiological cultures and hospitalizations that have been required.
Evaluate the number of patients who have required any of the bone or soft tissue reconstruction strategies. | Month 12
  Total number of new surgeries for better bone or soft tissue coverage: number of vacuum therapies (VAC or PICO), total number of grafts or flaps needed by the patient throughout the study.
Presentation of adverse events (frequency and severity). | Through study completion (12 months)
  Number of adverse events (frequency and severity) that have happened during the study.
Clostridium difficile infection | During treatment or 30 days after completion
  Number of cases observed during antibiotic treatment or 30 days after completion.

CONTACTS AND LOCATIONS:
Overall Officials: María Dolores del Toro López, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (29):
- Spain (29):
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Universitario El Bierzo, Ponferrada, León
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Virgen del Rocío, Seville, Seville
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Puerto Real, Cadiz
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Costa del Sol, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garrigos C, Rosso-Fernandez CM, Borreguero I, Rodriguez P, Garcia-Albea R, Bravo-Ferrer JM, Rodriguez-Bano J, Del Toro MD; DURATIOM team. Efficacy and safety of different antimicrobial DURATions for the treatment of Infections associated with Osteosynthesis Material implanted after long bone fractures (DURATIOM): Protocol for a randomized, pragmatic trial. PLoS One. 2023 May 22;18(5):e0286094. doi: 10.1371/journal.pone.0286094. eCollection 2023. PMID 37216357

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT05294796/SAP_000.pdf